CLINICAL TRIAL: NCT01920841
Title: A Blinded Comparison Trial of Two Topical Creams to Reduce Thigh Girth and to Smooth Thigh Skin in Women.
Acronym: ThighCream
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Design changed and will be resubmitted as a new study
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Nerium Biotechnology Inc (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2013-058
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Weight Loss
Keywords: lipolytic; herbal extracts; thigh girth; thigh smoothness
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left (A), Right (B) (Experimental): Cream A applied to left thigh and Cream B to right thigh
  Interventions: Other: Cream A applied to left thigh and Cream B to right thigh
- Left (B) Right (A) (Experimental): Cream B applied to left thigh and Cream A to right thigh
  Interventions: Other: Cream B applied to left thigh and Cream A to right thigh

INTERVENTIONS:
Other: Cream A applied to left thigh and Cream B to right thigh — Half the participants will receive Cream A applied to the left thigh, and Cream B applied to the right thigh
  Arms: Left (A), Right (B)
Other: Cream B applied to left thigh and Cream A to right thigh — Half the participants will receive Cream B applied to the left thigh and Cream A applied to the right thigh
  Arms: Left (B) Right (A)

SUMMARY:
The purpose of this study is to evaluate efficacy of two lipolytic creams differing in their bases and demonstrate that their herbal ingredients can reduce the size of the thigh and smooth the appearance of the thigh skin. It is hypothesized that creams with two different cream bases containing herbal products that stimulate the lipolytic process through stimulation of the beta-adrenergic receptor, with one cream base applied to each thigh daily 5 days a week for 4 weeks will reduce thigh girth and smooth the thigh skin compared to baseline.

DETAILED DESCRIPTION:
Participants will apply one cream (A) to one thigh and the second cream (B) to the other thigh under the supervision of a female clinic staff. The thigh to which each cream will be applied will be selected randomly, but half of the subjects will have cream A on the right thigh and cream B on the opposite thigh while the other half of the subjects will have the sides reversed. To evaluate the primary endpoint, both thighs will be measured at baseline and at the end of each treatment week, and the secondary endpoint will be assessed with standardized pictures of each thigh at baseline and on the last day of the fourth week which will end the study.

ELIGIBILITY:
Inclusion Criteria:

* Women who feel that their thighs are too large and the skin is insufficiently smooth.

Exclusion Criteria:

* Pregnant or nursing

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference in girth of the two thighs from baseline over the course of the treatment period | Four weeks
  Creams with two different cream bases containing forskolin, nerium oleander, salicin,caffeine, and green tea extract that have been shown to be safe topically will be evaluated. Both cream bases will be applied to the thighs daily 5 days a week for 4 weeks, with each thigh receiving the same cream base everyday. The thighs will be measured weekly

SECONDARY OUTCOMES:
Smoothness of the skin on the thighs treated with the two lipolytic creams differing in their bases compared to baseline using standardized photographs at baseline and at the end of the treatment. | Four weeks
  The secondary endpoint will be assessed with standardized pictures of each thigh at baseline and on the last day of the fourth week which will end the study.
Adverse events | 4 weeks
  Any adverse reaction to the creams will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States